CLINICAL TRIAL: NCT04871178
Title: Effects of a Mindfulness-Based Intervention on Symptoms and Signs, Well-Being and Health in Patients With Chronic Heart Failure
Brief Title: Dissertation Project Title: Effects of a Mindfulness-Based Intervention in Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro Ethical Sweden Dnr 265 10
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Chronic Heart Failure
Keywords: Feasibility study; Mindfulness interventions; Fatigue; Anxiety; Depression; Psychological Distress; Well-being; Health; Sense of coherence; Sleep; Dyspnea; Shortness of Breath; Breathlessness; Patient-reported outcomes
MeSH Terms: conditions — Fatigue; Anxiety Disorders; Depression; Dyspnea

STUDY DESIGN:
Intervention Model Description: A two-armed randomized, 8-week interventional and controlled (no intervention) feasibility study with two visits, one visit before (week 0) and one visit after intervention (week 10±1), with repeated measures
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Care as usual: (i.e. best medical treatment)
- Mindfulness-Based Intervention (Experimental): Care as usual (i.e. best medical treatment) in combination with an eight-week mindfulness-based educational and training program.
  Interventions: Behavioral: Mindfulness-based intervention

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — Eight, 2-hour instructor-led MBI group sessions once a week for 8 weeks, combined with formal meditative training at home for 20 minutes per day, 6 days a week.
  Course material consists of facts booklet, weekly training manuals, audio recordings on a CD, with the five formal guided meditative exercises (body scan, breathing anchor, breathing space, mindful movements, sitting meditation).
  The weekly home-work also included informal training of being present in daily life activities.
  The program is provided according to the standard MBI protocol. Compared to MBSR and MBCT durations of formal meditative practices are shorter and no 'all-day in silence' session is included. Because of participants' physical limitations and safety, the 'mindful movements' sequence, is adapted and performed in a sitting position.
  Adherence to the MBI was followed by self-reported weekly training in manuals asked to be submitted at group sessions.
  Other Names: MBI
  Arms: Mindfulness-Based Intervention

SUMMARY:
Patients with Chronic Heart Failure diagnosed and conventional treated, but still symptomatic (i.e. breathlessness, fatigue) is invited.

Eligible patients are randomised to (1) care as usual (i.e. optimized medical treatment) or (2) care as usual (i.e. optimized medical treatment) in combination with an 8-week mindfulness-based educational and training program.

Specific research questions:

* How are self-reported symptoms of breathlessness, fatigue, difficult sleeping, anxiety and depression affected by a mindfulness-based educational and training program (MBI)?
* Does the implementation of an 8-week Mindfulness-based program have any impact on personal experiences of well-being and health?
* What effects does an 8-week MBI have on objective signs of importance for the progression of heart failure?

DETAILED DESCRIPTION:
Effects of a Mindfulness-Based Intervention on Symptoms and Signs, Well-Being and Health in Patients with Chronic Heart Failure

Rationale: Despite progress in medical treatment, many patients with heart failure, still suffers from limiting symptoms with negative impact on their prognosis, wellbeing and health. Psychological distress, including anxiety and depression, is prevalent and difficult to treat in heart failure. Mindfulness-based interventions (MBIs), have shown beneficial effects on psychological and physiological symptoms, health and quality of life in other chronic conditions. The aims of the project were therefore to explore the feasibility and effects of MBI on symptoms and signs, well-being and health in patients diagnosed with chronic heart failure.

Hypothesis: was that outpatients with chronic heart failure would benefit from participating in an 8-week Mindfulness-based educational and training program (MBI) in addition to usual care (comprising standard health care and optimized medical treatment). With respect to (1) alleviate impact of symptoms (fatigue, breathlessness, impaired sleep, anxiety and depression), and (2) improve perceived wellbeing and health, and the sense of coherence (patient-reported outcomes), and (3) objective signs of importance for heart failure progression (heart rate, breathing rate, functional classification and capacity).

Study design: A prospective study, with a two-armed randomized and controlled designed, including two visits, was planned and initiated, integrated within the framework of a part-financed dissertation project. Complemented with qualitative research on participants' experiences of health, symptoms and the MBI.

Intervention: The intervention group received an 8-week MBI program in addition to treatment and care as usual (UC+MBI), while the control group received only treatment and care as usual (UC).

Data is collected in interviews and with clinical measurement of signs on site, and with validated patient-reported questionnaires, before and after 8-week intervention (UC+MBI) / Control (UC) period. Interviews were recorded and coded. Participants receive a minor physical examination with measurements of blood pressure, heart rate, breathing rate, weight and height, and assessment with a six-minute walk test. Participants is also provided with questionnaires to be answered at home, and send in to the University.

Nature and extend of the burden and risks: Due to the character of the MBI, with focused attention on thoughts, feelings and bodily sensations, emotional reactions may be a risk (as is described in Informed Consent Form). Participants were free to contact with the MBI instructor or a counsellor, during study period. The burden of participation (i.e. time investment in learning the mindfulness-based meditative training and extra study examinations) may be compensated by the possible benefits.

The present study has been carried through within the framework of a part-financed dissertation project with four sub-projects. The feasibility study, showing patients recruitment and flow through the study, with results of the MBI on symptoms and signs in patients with chronic heart failure is published [1].

The study has not prior been registered at clinicalTrial.gov, due to the nature of the interventional pilot study, as was original initiated as a part of a Master Thesis, and registration was not required at the time recruitment began in 2010. Also, it is not until now we realize the value to retrospectively register the study, when able to provide the new knowledge gained by the project in the sub-project II, III and IV.

The study has been conducted in several phases, including a pre-pilot phase and two pilot phases. In the pre-pilot phase, the study protocol with the Research Person Information (Informed Consent Form) was evaluated with patients randomly assigned to a MBI (n=3) or control group (n=3). Results on participants' experiences of the MBI, and the effects on the outcomes, were analyzed with a qualitative approach and described in a Master's thesis (in Swedish).

The present study protocol was approved in 2010, by the Regional Ethical Board in Gothenburg, Sweden (No. 265:10), with a few minor revisions, including tuning down the benefits, and the advice to review if possible, to reduce the number of instruments in the study.

All through the study has been performed according to the principles of the Declaration of Helsinki. All participants provided written and Informed Consent and signed the ICF before beginning the study, and were informed of the right of free withdrawal.

The first pilot phase lasted from 2010 to 2011. In February 2012 the study was approved for a doctoral student position, with research grants from the Centre for Person-Centred Care at the University of Gothenburg (GPCC). GPCC was founded by the Swedish Government´s grant for Strategic Research Areas, Care Sciences (Application to Swedish Council no. 2009-1088). The second phase of the study was conducted in 2013, called the "Main study", but the RCT was to be transformed to a feasibility study.

The Analysis plan into the dissertation project: Effects of a Mindfulness-Based Intervention on Symptoms and Signs, Well-being and Health in patients with Chronic Heart Failure, includes both qualitative and quantitative methods. Briefly, the original focus on qualitative research, shifted to emphasis quantitative methods. The original plan to use parametric methods, to compare the study groups, shifted to Non-parametric Mann-Whitney U test. Due to the small sample size, and the ordinal level of data. Statistical analysis was carried out in consultation with Healthmetrics, University of Gothenburg, Sweden. Two separate sets of outcome variables were constructed prior analysis. The first set was on symptoms and signs and included in published paper [1]. The other set is on the psychological outcomes (anxiety and depression), well-being, sense of coherence and health [paper II). Paper III is a qualitative: Experiences of Breathing and Shortness of Breath with Chronic Heart Failure - A descriptive and explorative study. The 4th paper is a Mixed-Method study on the effects of MBI on problematic shortness of breath experiences with heart failure.

Topics of research in this project may be relevant for many patients with heart failure and professionals. The reasons for delay of publishing results in the present study is several, what matters now is the ability to share the new knowledge on the effects of MBI on psychological distress and health in heart failure with patients and professionals all over the world. That is the heart goal for this application to ClinicalTrial.gov.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed chronic heart (CHF) failure by echocardiography
* Functional class II-IV according to the New York Heart Association (NYHA)
* Symptoms of breathlessness and/or tiredness rated 2-5 by patients using five-point scales, ranging from asymptomatic (1) to symptoms at rest (5)
* Stable condition, that is no deterioration of heart failure symptoms or new CHF drug or hospitalizations because of decompensated heart failure within the last four weeks

Exclusion Criteria:

* Severe psychiatric diagnosis (requiring treatment)
* Severe substance abuse (documented in journal)
* Severe somatic disease with short expected survival (i.e., malignancy)
* Communication difficulties (i.e., impaired vision or hearing, need of an interpreter to understand Swedish)
* Cognitive or adherence difficulties (documented in journal)
* Unstable angina pectoris
* Post-partum cardiomyopathy
* Ongoing participation in any other interventional study
* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10-10 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Self-reported impact of fatigue | 10 weeks
  Change from baseline to follow-up at week 10, will be measured at the Fatigue Severity Scale (FSS), a self-administered questionnaire including nine items investigating the impact of disabling fatigue on daily functioning during the past week. Grading of each item ranges from 1 to 7, with the total possible fatigue sum score ranging from 9 to 63, and higher scores indicating higher levels of indexed impact of fatigue. The FSS had not previously been tested in a heart failure population, and no cut-off score was found. The FSS was provided at visits and answered at home, and sent in to University address.

SECONDARY OUTCOMES:
Anxiety | 10 weeks
  Change from baseline to follow-up at week 10, will be measured at the Hospital Anxiety and Depression Scale (HADS). The HADS is a self-administered questionnaire with two sub-scales to detect possible presence of anxiety (HADS-A) and/or depression (HADS-D). Both sub-scales include 7 items, with four-point scales ranging from 0 to 3, with total sum-score ranging from 0-21, and defined as 0-7 (normal), 8-10 (possible case), and 11-21 (probable case) of anxiety disorders or depression, and the patient in need of additional psychiatric treatment. Optimal cut-off for both subscales is set to ≥8. The HADS was provided at visits, answered at home, and sent to University address.
Depression | 10 weeks
  Change from baseline to follow-up at week 10, will be measured at the Hospital Anxiety and Depression Scale (HADS). The HADS is a self-administered questionnaire with two sub-scales to detect possible presence of anxiety (HADS-A) and/or depression (HADS-D). Both sub-scales include 7 items, with four-point scales ranging from 0 to 3, with total sum-score ranging from 0-21, and defined as 0-7 (normal), 8-10 (possible case), and 11-21 (probable case) of anxiety disorders or depression, and the patient in need of additional psychiatric treatment. Optimal cut-off for both subscales is set to ≥8. The HADS was provided at visits, answered at home, and sent to University address.
Psychological and General Well-Being | 10 weeks
  Change from baseline to follow-up at week 10, will be measured at the Psychological and General Well-Being (PGWB) index. The PGWB is a 22-item self-administered questionnaire designed to measure "self-representations of intrapersonal affective or emotional states reflecting a sense of subjective well-being or distress. The six response options were coded 1-6 in accordance with Swedish studies, and the total PGWB sum score was ranging from 22 to 132, with defined categories (1) score 22-82 (Severe distress); (2) score 83-94 (Moderate distress); score 95-132 (Positive well-being). The PGWB was provided at visits, answered at home, and sent in to University address.
Sense of coherence | 10 weeks
  Change from baseline to follow-up at week 10, will be measured at the self-administered questionnaire Sense of coherence (SOC-13) total index. The SOC-13 consisting of 13 items, all with seven-point scale and two anchoring responses. With higher scores indicating higher personal capabilities to perceive the world and stressful events in life as comprehensible, manageable, and meaningful defined as high SOC. The psychometric tested Swedish version of SOC-13, and the total score categories defined as: 30-60 (Low SOC); 61-75 (Moderate SOC); 76-91 (High SOC) is used. The SOC-13 was provided at visits, answered at home, and sent in to University address.
Health | 10 weeks
  Change from baseline to follow-up at week 10, on self-reported health, will be measured at the Swedish version of the 36-item Short Form Health Survey (SF-36) General Health (GH) Index. The SF-36 GH index consists of five items, with questions focusing participants' perception of their health, with five response choices each, and higher points indicating better health. The SF-36 questionnaire were included in the first phase (pilot 1), then temporary removed. The value of health status as measured in the SF-36, was reconsidered 2012 and the instrument was reinstated in 2013 (pilot 2). The SF-36 was provided at visits, answered at home, and sent in to University address.
Self-reported symptoms of impaired sleep | 10 weeks
  Change from baseline to follow-up at week 10, will be measured at the Karolinska Sleep Questionnaire - sleep quality index (KSQ-sqi). Which is a sub-scale including four questions, with high scores indicating good sleep quality. The KSQ was provided at visits, answered at home, and sent to University address.

OTHER OUTCOMES:
Heart rate | 10 weeks
  Change from baseline to follow-up at week 10, in heart rate (beats/min), will be measured in sitting position after rest (>5 min) using an automated non-invasive monitor (Omron Memory Intelli Sense, model 705 IT; Omron Healthcare, Hoofddorp, The Netherlands). With a lower heart rate frequency representing a better prognostic sign.
Respiratory rate | 10 weeks
  Change from baseline to follow-up at week 10, in respiratory rate, will be assessed manually using the pulse clock, at rest within a set of 60 s. With a calmer breathing rate representing a better sign, and higher rates to be a worsening heart failure sign, as linked to fluid retention in the body and decompensation.
Functional classification | 10 weeks
  Change from baseline to follow-up at week 10, in New York Heart Association (NYHA class). With the NYHA class based on patient-reported symptoms on five-point Likert scale (breathlessness and tiredness) as related to physical exertion. Patient response alternatives ranged from (1) 'I am never breathless/tired' to (5) 'when I am at rest', with each symptom reported separately. With a lower NYHA class indicating lower severity degree of symptoms and improved physical function.
Breathlessness related to physical exertion | 10 weeks
  Change from baseline to follow-up at week 10, in the patient-reported severity of breathlessness related to physical activity, using five-point Likert scale. Patients' response alternatives ranged from: (1) asymptomatic 'I am never breathless'; (2) 'When I am walking up the stairs (one floor) or in a slope at normal pace'; (3) 'Walking at normal pace on a flat surface (< 200 m)'; (4) 'Walking slowly on flat surface (< 100 m) or during washing or dressing'; up to (5) 'When I am at rest'.
Tiredness related to physical exertion | 10 weeks
  Change from baseline to follow-up at week 10, in the patient-reported severity of tiredness, related to physical activity, using five-point Likert scale. Patients' response alternatives ranged from (1) asymptomatic 'I am never tired'; (2) 'When I am walking up the stairs (one floor) or in a slope at normal pace'; (3) 'Walking at normal pace on a flat surface (< 200 m)'; (4) 'Walking slowly on flat surface (< 100 m) or during washing or dressing'; up to (5) ('When I am at rest').
Functional capacity | 10 weeks
  Change from baseline to follow-up at week 10, measured in distance (in meter) walked at the 6-min walk test. With a longer distance walked in 6 minutes, indicating improved functional capacity. Additional outcome assessed as 'objective sign', in participants in the second phase of the study.
Shortness of breath | 10 weeks
  Change from baseline to follow-up at week 10, will be measured and described in self-reported experiences of breathing and shortness of breath explored in semi structured interviews, guided by an extended assessment tool "Experiences of Breathing and Shortness of breath" (Exp-BeSoB), in development within the project. The Exp-BeSoB includes both open-ended questions, where participants are allowed to explore their own experiences in several dimensions, and pre-formulated descriptors, and self-rating scales related to shortness of breath experiences. With lower scores indicating alleviated breathing symptoms.
Other symptoms | 10 weeks
  Change from baseline to follow-up at week 10, will be measured in six other self-reported symptoms (ankle swelling, impaired appetite; nausea, pain at rest/moving, thirst/dryness in the throat, and unsteadiness/dizziness) commonly reported by patients with chronic heart failure. Occurrence of symptom within a timeframe of "last week" ("no/yes"), and the degree of symptom severity self-reported by participants using 11-point numerical rating scale (NRS) ranging from 0 ("not at all bothersome") to 10 ("worst possible"), with higher rating degree indicating more severe symptom experiences.
Health self-rated on Visual Analogue Scale | 10 weeks
  Change from baseline to follow-up at week 10, in health will be measured using self-rating scales. In the first pilot (2010 - 2011) health was also assessed on an ungraded vertical visual analog scale (VAS), with the anchor points "worse health" and "best health" (at the top of the scale). The scale was in 2013, changed into a horizontal 11-point numerical rating scale (NRS) ranging from 0 ("worst possible health") to 10 ("best possible health"). Due to different scale measures, outcome was not possible to include in statistical analysis. Health measures on VAS were used in the 2nd sub-project to identify outliers among participants who didn't answer the SF-36, in the first pilot.
Well-being self-rated on Likert-scale | 10 weeks
  Change from baseline to follow-up at week 10, in well-being as measured on self-rating scales. In the first pilot (2010 - 2011) well-being was also assessed on a 5-point Likert scale (1-5), with the anchor points (1) "no well-being" and (5) "best possible well-being". The scale was in 2013, also changed into a horizontal 11-point numerical rating scale (NRS) ranging from 0 to 10 with the anchor points (1) "worst possible well-being" and (10) "best possible well-being". Due to different scale measures, outcome was not possible to include in statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lena M Björck Associate Professor, PhD, RN, Principal Investigator — Göteborg University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Paren P, Schaufelberger M, Bjorck L, Lappas G, Fu M, Rosengren A. Trends in prevalence from 1990 to 2007 of patients hospitalized with heart failure in Sweden. Eur J Heart Fail. 2014 Jul;16(7):737-42. doi: 10.1002/ejhf.109. Epub 2014 May 26. PMID 24863749
- [Background] Zambroski CH, Moser DK, Bhat G, Ziegler C. Impact of symptom prevalence and symptom burden on quality of life in patients with heart failure. Eur J Cardiovasc Nurs. 2005 Sep;4(3):198-206. doi: 10.1016/j.ejcnurse.2005.03.010. PMID 15916924
- [Background] Barnes S, Gott M, Payne S, Parker C, Seamark D, Gariballa S, Small N. Prevalence of symptoms in a community-based sample of heart failure patients. J Pain Symptom Manage. 2006 Sep;32(3):208-16. doi: 10.1016/j.jpainsymman.2006.04.005. PMID 16939845
- [Background] Falk K, Swedberg K, Gaston-Johansson F, Ekman I. Fatigue is a prevalent and severe symptom associated with uncertainty and sense of coherence in patients with chronic heart failure. Eur J Cardiovasc Nurs. 2007 Jun;6(2):99-104. doi: 10.1016/j.ejcnurse.2006.05.004. Epub 2006 Jul 10. PMID 16831569
- [Background] Janssen DJ, Spruit MA, Uszko-Lencer NH, Schols JM, Wouters EF. Symptoms, comorbidities, and health care in advanced chronic obstructive pulmonary disease or chronic heart failure. J Palliat Med. 2011 Jun;14(6):735-43. doi: 10.1089/jpm.2010.0479. Epub 2011 Apr 21. PMID 21510771
- [Background] Yohannes AM, Willgoss TG, Baldwin RC, Connolly MJ. Depression and anxiety in chronic heart failure and chronic obstructive pulmonary disease: prevalence, relevance, clinical implications and management principles. Int J Geriatr Psychiatry. 2010 Dec;25(12):1209-21. doi: 10.1002/gps.2463. PMID 20033905
- [Background] Wu JR, Lennie TA, Frazier SK, Moser DK. Health-Related Quality of Life, Functional Status, and Cardiac Event-Free Survival in Patients With Heart Failure. J Cardiovasc Nurs. 2016 May-Jun;31(3):236-44. doi: 10.1097/JCN.0000000000000248. PMID 25774841
- [Background] Steptoe A, Mohabir A, Mahon NG, McKenna WJ. Health related quality of life and psychological wellbeing in patients with dilated cardiomyopathy. Heart. 2000 Jun;83(6):645-50. doi: 10.1136/heart.83.6.645. PMID 10814621
- [Background] Falk K, Granger BB, Swedberg K, Ekman I. Breaking the vicious circle of fatigue in patients with chronic heart failure. Qual Health Res. 2007 Oct;17(8):1020-7. doi: 10.1177/1049732307306914. PMID 17928476
- [Background] Ekman I, Kjellstrom B, Falk K, Norman J, Swedberg K. Impact of device-guided slow breathing on symptoms of chronic heart failure: a randomized, controlled feasibility study. Eur J Heart Fail. 2011 Sep;13(9):1000-5. doi: 10.1093/eurjhf/hfr090. Epub 2011 Jul 28. PMID 21803755
- [Background] Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. J Behav Med. 1985 Jun;8(2):163-90. doi: 10.1007/BF00845519. PMID 3897551
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Sundquist J, Lilja A, Palmer K, Memon AA, Wang X, Johansson LM, Sundquist K. Mindfulness group therapy in primary care patients with depression, anxiety and stress and adjustment disorders: randomised controlled trial. Br J Psychiatry. 2015 Feb;206(2):128-35. doi: 10.1192/bjp.bp.114.150243. Epub 2014 Nov 27. PMID 25431430
- [Background] Sundquist J, Palmer K, Johansson LM, Sundquist K. The effect of mindfulness group therapy on a broad range of psychiatric symptoms: A randomised controlled trial in primary health care. Eur Psychiatry. 2017 Jun;43:19-27. doi: 10.1016/j.eurpsy.2017.01.328. Epub 2017 Feb 8. PMID 28365464
- [Background] Kenne Sarenmalm E, Martensson LB, Andersson BA, Karlsson P, Bergh I. Mindfulness and its efficacy for psychological and biological responses in women with breast cancer. Cancer Med. 2017 May;6(5):1108-1122. doi: 10.1002/cam4.1052. Epub 2017 Apr 18. PMID 28421677
- [Background] Sundquist J, Palmer K, Memon AA, Wang X, Johansson LM, Sundquist K. Long-term improvements after mindfulness-based group therapy of depression, anxiety and stress and adjustment disorders: A randomized controlled trial. Early Interv Psychiatry. 2019 Aug;13(4):943-952. doi: 10.1111/eip.12715. Epub 2018 Jul 3. PMID 29968371
- [Background] Saha S, Jarl J, Gerdtham UG, Sundquist K, Sundquist J. Economic evaluation of mindfulness group therapy for patients with depression, anxiety, stress and adjustment disorders compared with treatment as usual. Br J Psychiatry. 2020 Apr;216(4):197-203. doi: 10.1192/bjp.2018.247. PMID 30468136
- [Background] Sullivan MJ, Wood L, Terry J, Brantley J, Charles A, McGee V, Johnson D, Krucoff MW, Rosenberg B, Bosworth HB, Adams K, Cuffe MS. The Support, Education, and Research in Chronic Heart Failure Study (SEARCH): a mindfulness-based psychoeducational intervention improves depression and clinical symptoms in patients with chronic heart failure. Am Heart J. 2009 Jan;157(1):84-90. doi: 10.1016/j.ahj.2008.08.033. PMID 19081401
- [Background] Viveiros J, Chamberlain B, O'Hare A, Sethares KA. Meditation interventions among heart failure patients: An integrative review. Eur J Cardiovasc Nurs. 2019 Dec;18(8):720-728. doi: 10.1177/1474515119863181. Epub 2019 Jul 23. PMID 31331192
- [Background] Scott-Sheldon LAJ, Gathright EC, Donahue ML, Balletto B, Feulner MM, DeCosta J, Cruess DG, Wing RR, Carey MP, Salmoirago-Blotcher E. Mindfulness-Based Interventions for Adults with Cardiovascular Disease: A Systematic Review and Meta-Analysis. Ann Behav Med. 2020 Jan 1;54(1):67-73. doi: 10.1093/abm/kaz020. PMID 31167026
- [Background] RICKHAM PP. HUMAN EXPERIMENTATION. CODE OF ETHICS OF THE WORLD MEDICAL ASSOCIATION. DECLARATION OF HELSINKI. Br Med J. 1964 Jul 18;2(5402):177. doi: 10.1136/bmj.2.5402.177. No abstract available. PMID 14150898
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Dupuy HJ. The Psychological General Well-Being (PGWB) Index. New York: Le Jacq; 1984
- [Background] Antonovsky A. The structure and properties of the sense of coherence scale. Soc Sci Med. 1993 Mar;36(6):725-33. doi: 10.1016/0277-9536(93)90033-z. PMID 8480217
- [Background] Langius A, Bjorvell H, Antonovsky A. The sense of coherence concept and its relation to personality traits in Swedish samples. Scand J Caring Sci. 1992;6(3):165-71. doi: 10.1111/j.1471-6712.1992.tb00146.x. PMID 1439378
- [Background] Sullivan M, Karlsson J, Ware JE Jr. The Swedish SF-36 Health Survey--I. Evaluation of data quality, scaling assumptions, reliability and construct validity across general populations in Sweden. Soc Sci Med. 1995 Nov;41(10):1349-58. doi: 10.1016/0277-9536(95)00125-q. PMID 8560302
- [Background] Sullivan M, Karlsson J. The Swedish SF-36 Health Survey III. Evaluation of criterion-based validity: results from normative population. J Clin Epidemiol. 1998 Nov;51(11):1105-13. doi: 10.1016/s0895-4356(98)00102-4. PMID 9817128
- [Background] Ware JE, Kosinski M. Interpreting SF-36 summary health measures: a response. Qual Life Res. 2001;10(5):405-13; discussion 415-20. doi: 10.1023/a:1012588218728. PMID 11763203
- [Background] Kecklund G, Akerstedt T. The psychometric properties of the Karolinska Sleep Questionnaire. J Sleep Res 1992;6:221-29.
- [Background] Bennett JA, Riegel B, Bittner V, Nichols J. Validity and reliability of the NYHA classes for measuring research outcomes in patients with cardiac disease. Heart Lung. 2002 Jul-Aug;31(4):262-70. doi: 10.1067/mhl.2002.124554. PMID 12122390
- [Background] Ekman I, Cleland JG, Swedberg K, Charlesworth A, Metra M, Poole-Wilson PA. Symptoms in patients with heart failure are prognostic predictors: insights from COMET. J Card Fail. 2005 May;11(4):288-92. doi: 10.1016/j.cardfail.2005.03.007. PMID 15880338
- [Background] Vuckovic KM, Fink AM. The 6-min walk test: is it an effective method for evaluating heart failure therapies? Biol Res Nurs. 2012 Apr;14(2):147-59. doi: 10.1177/1099800411403918. Epub 2011 May 17. PMID 21586495
- [Background] Ekman I, Granger B, Swedberg K, Stenlund H, Boman K. Measuring shortness of breath in heart failure (SOB-HF): development and validation of a new dyspnoea assessment tool. Eur J Heart Fail. 2011 Aug;13(8):838-45. doi: 10.1093/eurjhf/hfr062. PMID 21791539
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Krippendorf K. Content analysis. An introduction to its methodology. 6th ed. London: Sage; 2004.
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Janson Fagring A, Gaston-Johansson F, Danielson E. Description of unexplained chest pain and its influence on daily life in men and women. Eur J Cardiovasc Nurs. 2005 Dec;4(4):337-44. doi: 10.1016/j.ejcnurse.2005.06.003. Epub 2005 Nov 10. PMID 16289921
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Meleis AI, Sawyer LM, Im EO, Hilfinger Messias DK, Schumacher K. Experiencing transitions: an emerging middle-range theory. ANS Adv Nurs Sci. 2000 Sep;23(1):12-28. doi: 10.1097/00012272-200009000-00006. PMID 10970036
- [Background] Meditation practice for health. State of research. Evidens report/technology assessment. Agency for healthcare research and quality. University of Alberta Evidence-based Practice Centre. Number 155, 2007,
- [Background] Arias AJ, Steinberg K, Banga A, Trestman RL. Systematic review of the efficacy of meditation techniques as treatments for medical illness. J Altern Complement Med. 2006 Oct;12(8):817-32. doi: 10.1089/acm.2006.12.817. PMID 17034289
- [Background] Chang BH, Hendricks A, Zhao Y, Rothendler JA, LoCastro JS, Slawsky MT. A relaxation response randomized trial on patients with chronic heart failure. J Cardiopulm Rehabil. 2005 May-Jun;25(3):149-57. doi: 10.1097/00008483-200505000-00005. PMID 15931018
- [Background] Curiati JA, Bocchi E, Freire JO, Arantes AC, Braga M, Garcia Y, Guimaraes G, Fo WJ. Meditation reduces sympathetic activation and improves the quality of life in elderly patients with optimally treated heart failure: a prospective randomized study. J Altern Complement Med. 2005 Jun;11(3):465-72. doi: 10.1089/acm.2005.11.465. PMID 15992231
- [Background] Bernardi L, Spadacini G, Bellwon J, Hajric R, Roskamm H, Frey AW. Effect of breathing rate on oxygen saturation and exercise performance in chronic heart failure. Lancet. 1998 May 2;351(9112):1308-11. doi: 10.1016/S0140-6736(97)10341-5. PMID 9643792
- [Background] Baer RA, Mindfulness Training as a clinical intervention: A Conceptual and Emperical Review. Clin Psychol Sci Prac 2003;10(2):125-143.
- [Background] Davidson RJ, Kabat-Zinn J, Schumacher J, Rosenkranz M, Muller D, Santorelli SF, Urbanowski F, Harrington A, Bonus K, Sheridan JF. Alterations in brain and immune function produced by mindfulness meditation. Psychosom Med. 2003 Jul-Aug;65(4):564-70. doi: 10.1097/01.psy.0000077505.67574.e3. PMID 12883106
- [Background] Hirshberg MJ, Goldberg SB, Rosenkranz M, Davidson RJ. Prevalence of harm in mindfulness-based stress reduction. Psychol Med. 2022 Apr;52(6):1080-1088. doi: 10.1017/S0033291720002834. Epub 2020 Aug 18. PMID 32807249
- [Background] Levine GN, Lange RA, Bairey-Merz CN, Davidson RJ, Jamerson K, Mehta PK, Michos ED, Norris K, Ray IB, Saban KL, Shah T, Stein R, Smith SC Jr; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; and Council on Hypertension. Meditation and Cardiovascular Risk Reduction: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2017 Sep 28;6(10):e002218. doi: 10.1161/JAHA.117.002218. PMID 28963100
- [Background] Krittanawong C, Kumar A, Wang Z, Narasimhan B, Jneid H, Virani SS, Levine GN. Meditation and Cardiovascular Health in the US. Am J Cardiol. 2020 Sep 15;131:23-26. doi: 10.1016/j.amjcard.2020.06.043. Epub 2020 Jun 30. PMID 32758360
- [Background] Jaarsma T, Hill L, Bayes-Genis A, La Rocca HB, Castiello T, Celutkiene J, Marques-Sule E, Plymen CM, Piper SE, Riegel B, Rutten FH, Ben Gal T, Bauersachs J, Coats AJS, Chioncel O, Lopatin Y, Lund LH, Lainscak M, Moura B, Mullens W, Piepoli MF, Rosano G, Seferovic P, Stromberg A. Self-care of heart failure patients: practical management recommendations from the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2021 Jan;23(1):157-174. doi: 10.1002/ejhf.2008. Epub 2020 Oct 20. PMID 32945600
- [Background] Heidenreich PA, Fonarow GC, Breathett K, Jurgens CY, Pisani BA, Pozehl BJ, Spertus JA, Taylor KG, Thibodeau JT, Yancy CW, Ziaeian B. 2020 ACC/AHA Clinical Performance and Quality Measures for Adults With Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Performance Measures. J Am Coll Cardiol. 2020 Nov 24;76(21):2527-2564. doi: 10.1016/j.jacc.2020.07.023. Epub 2020 Nov 2. No abstract available. PMID 33153861
- [Background] Schenström O. (in Swedish) (2007) Mindfulness i vardagen - vägar till medveten närvaro. 10th edition Viva Publishing House by Ljungbergs sätteri i Köping, printed 2009 by ScandBook AB in Falun, Sweden.
- [Background] Schenström O. (in Swedish) Här & Nu - Ett program för medveten närvaro; 2013. The MBI program is available from web site: http://www.mindfulnesscenter.se Accessed April 15, 2021, but is not linked due to the site also includes other mindfulness-based educational program, products and services.
- [Result] Norman J, Fu M, Ekman I, Bjorck L, Falk K. Effects of a mindfulness-based intervention on symptoms and signs in chronic heart failure: A feasibility study. Eur J Cardiovasc Nurs. 2018 Jan;17(1):54-65. doi: 10.1177/1474515117715843. Epub 2017 Jun 22. PMID 28639841